CLINICAL TRIAL: NCT06025539
Title: Effects of an Animal-assisted Resilience Training for Children With a History of Stressful Life Events or a Diagnosis of Autism Spectrum Disorder: A Pilot Study
Brief Title: Animal-assisted Resilience Training for Children With Stressful Life Events or Autism Spectrum Disorder
Acronym: AART
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Resilience training
Record Dates: First submitted 2023-08-22; First posted 2023-09-06 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder; Life Change Events
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Animal-assisted resilience training (Experimental): 12 sessions of group-based, animal-assisted resilience training.
  Interventions: Behavioral: Animal-assisted resilience training

INTERVENTIONS:
Behavioral: Animal-assisted resilience training — Participants take part in 12 sessions (120 minutes each), each session focuses on a topic that is related to resilience. The intervention takes part outdoors on a farm, and includes interactions with several different animals. The training takes place in small groups, and includes exercises, observations, and discussions.

SUMMARY:
The goal of this clinical trial is to learn about the effects of an animal-assisted resilience training in children who experienced stressful life events or who have a diagnosis of autism spectrum disorder. The main question it aims to answer is:

• Is an animal-assisted resilience training a feasible approach to increase resilience in children with a history of stressful life events or a diagnosis of autism spectrum disorder?

Participants will take part in 12 training sessions of a standardized resilience training. The training is group-based, takes place outdoors, and includes interactions with different animals. It focuses on self-esteem, self-perception, dealing with emotions, and social competence.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 and 4 years (toddler group) or 8 and 12 years (children group)
* History of at least one stressful life event experience OR diagnosis of autism spectrum disorder
* Basic knowledge of either German or English of parents and child to follow the instructions during the training sessions and completion of interviews.

Exclusion Criteria:

- Medical contraindications for contact with animals, such as allergies or phobia

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Questionnaire on resources in childhood and adolescence | 18 weeks
  Pre-to-post assessment changes in resilience

SECONDARY OUTCOMES:
Questionnaire to assess emotion regulation in children and adolescents | 18 weeks
  Pre-to-post assessment changes in emotion regulation
Number of attended sessions | 12 weeks
  Number of attended sessions over the course of the training
Feeling secure and motivation to participate as measured on a 0-10 scale | 12 weeks
  Motivation and feeling secure as measured at the beginning and end of each session
Intervention satisfaction as assessed in semi-structured interview | 18 weeks (follow-up)
  Satisfaction with program content and structure, as measured by qualitative interview
Strengths and Difficulties Questionnaire (SDQ) | 18 weeks
  Pre-to-post assessment changes in peer-relationship problems and prosocial behavior measures

CONTACTS AND LOCATIONS:
Locations (1):
- University of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
Data will be shared upon request and only once study results have been published.